CLINICAL TRIAL: NCT04119037
Title: Percutaneous Cordotomy for Pain Palliation in Advanced Cancer
Brief Title: Cordotomy in Reducing Pain in Patients With Advanced Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2019-0264; NCI-2019-03708 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2019-0264 (Other: M D Anderson Cancer Center); R01NR018481 (NIH)
Record Dates: First submitted 2019-09-11; First posted 2019-10-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Advanced Malignant Neoplasm
MeSH Terms: interventions — Cordotomy; Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I (cordotomy) (Experimental): Patients undergo a cordotomy over 1-2 hours.
  Interventions: Procedure: Cordotomy; Other: Questionnaire Administration
- Group II (morphine, fake cordotomy) (Sham Comparator): Patients receive morphine via injection into the spine and undergo a fake cordotomy over 1-2 hours.
  Interventions: Drug: Morphine; Other: Questionnaire Administration; Procedure: Sham Intervention

INTERVENTIONS:
Procedure: Cordotomy — Undergo cordotomy
  Arms: Group I (cordotomy)
Drug: Morphine — Given via injection
  Arms: Group II (morphine, fake cordotomy)
Other: Questionnaire Administration — Ancillary studies
Procedure: Sham Intervention — Undergo fake cordotomy
  Arms: Group II (morphine, fake cordotomy)

SUMMARY:
This trial studies how well cordotomy works in reducing pain in patients with cancer that has spread to other places in the body (advanced). Cordotomy is performed on the spinal cord with a needle and guided by computed tomography scans and is designed to help reduce pain. This study is being done to learn if a cordotomy reduces pain in patients with unmanageable cancer pain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Assess the efficacy of cordotomy for patients with unilateral advanced cancer pain.

SECONDARY OBJECTIVES:

I. Define the patient experience of cordotomy for cancer pain refractory to palliative care.

II. Determine whether magnetic resonance imaging (MRI) can be used as a noninvasive biomarker for a successful cordotomy.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo a cordotomy over 1-2 hours.

GROUP II: Patients receive morphine via injection into the spine and undergo a fake cordotomy over 1-2 hours.

After completion of study, patients are followed up at 2 weeks and once every month for up to 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Has undergone 3 palliative care evaluations
* Pain intensity >= 4 on a 0-10 numerical scale
* Unilateral pain due to cancer below the shoulder level (arm, trunk, hip, leg)

Exclusion Criteria:

* Uncorrectable coagulopathy
* Large intracranial mass
* Inability to complete assessment forms
* Life expectancy < 1 month
* Contraindication to intravenous sedation
* Morphine allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-09-16 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in pain intensity | Up to 6 months
  Will be measured by the Edmonton Symptom Assessment Scale (ESAS).

SECONDARY OUTCOMES:
Brief Pain Inventory pain interference items | Up to 6 months
  Will provide initial estimates of the magnitude of the effect of cordotomy.
Other ESAS symptoms | Up to 6 months
  Will provide initial estimates of the magnitude of the effect of cordotomy.

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bruera, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org